CLINICAL TRIAL: NCT04295044
Title: Effect of High Protein Diet in Stroke Patients With Low Muscle Mass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORPG6G0191
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke; Diet, Healthy; Muscle Loss
MeSH Terms: conditions — Ischemic Stroke; Muscular Atrophy | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein diet (Experimental): received high protein diet, prescribed by dietitian
  Interventions: Dietary Supplement: high protein diet
- Normal protein diet (Active Comparator): received normal protein diet, prescribed by dietitian
  Interventions: Dietary Supplement: normal protein diet

INTERVENTIONS:
Dietary Supplement: high protein diet — receive 1.8g protein/kg
  Arms: High protein diet
Dietary Supplement: normal protein diet — receive 1g protein/kg
  Arms: Normal protein diet

SUMMARY:
Our prior studies demonstrated that dehydration was a predictor for poor outcome in stroke and Blood urea nitrogen/Cr ratio-based saline hydration therapy in patients with acute ischemic stroke may increase the rate of favorable clinical outcome with functional independence at 3 months after stroke. However, dehydration is likely to be only a part of representation in poor nutrition status and physical fragility for a stroke patient.

Our prior study found that acute stroke patients admitted to neurological intensive care unit with low urinary creatinine excretion rate (CER), a marker of muscle mass, was associated with poor outcome at 6 months after stroke. An animal study suggested inadequate food and water intake determine mortality following stroke in mice and nutritional support reduced the 14-day mortality rate from 59% to 15%. A study also showed that high protein intake was associated with a better outcome in previous cardiovascular events.

We will calculate CER based on published equation. Based on our prior study, acute stroke patients with their CER<1500 mg/day will be enrolled. A randomized controlled trial will be conducted and patients will be randomly assigned to high protein diet or normal protein diet for at least 2 weeks. We plan to enroll 300 patients, with 150 patients in ach group, during 3-year study period. We will consult dietitians for arrangement of their diet. We assume that patients receiving high protein diet will have higher opportunity to walk independently (modified Rankin Scale 0-1) at 3 month after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke during hospitalization
2. eGFR >30
3. urine albumin creatinine ratio < 30 mg/g
4. urinary creatinine excretion rate (CER) < 1500g/day

Exclusion Criteria:

1. chronic kidney disease stage 4 or 5 (i.e. eGFR < 30)
2. proteinuria (protein 1+ or more in urine routine)
3. known impairment of functional status (mRS ≥ 2) prior to the index stroke
4. refuse to participate in this study.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale 0-1 | 3 months
  No significant disability

SECONDARY OUTCOMES:
modified Rankin Scale 0-2 | 3 months
  Slight disability

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No